CLINICAL TRIAL: NCT02484664
Title: COLA: A Pilot Clinical Trial of COX-2 Inhibition in LAM and TSC
Acronym: COLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Kwiatkowski, Professor and Senior Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000954
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Results first posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Lymphangioleiomyomatosis (LAM)
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- celecoxib (Experimental): Celecoxib 200mg PO QD for 6 months
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — We will perform a pilot clinical trial to investigate the safety and tolerability of celecoxib therapy as a single agent for patients with LAM. LAM subjects who are not taking everolimus or rapamycin will be treated with celecoxib at 200mg PO QD for 6 months. They will be monitored for respiratory function and angiomyolipoma size. At the end of the 6 month period, celecoxib will be discontinued, and subjects will be monitored for another 6 months.

SUMMARY:
The investigators will perform a two-center phase I trial of celecoxib (COX-2 inhibitor) administered at 200mg by mouth daily for 6 months. Up to 12 adult women with LAM will be recruited (between 4-8 at each site). The Specific Aims are:

Aim 1: To investigate whether, in LAM patients, celecoxib is safe and well tolerated, and has evidence of clinical benefit.

Aim 2: To investigate the potential value of a novel biomarker of LAM, quantitative measurement of the number of TSC2 mutant LAM cells per ml of blood, to assess disease severity.

DETAILED DESCRIPTION:
Background: Lymphangioleiomyomatosis (LAM) is characterized by cystic lung destruction, kidney angiomyolipomas (AMLs), and LAM cell growth within the axial lymphatics and multiple other organs and surfaces. LAM occurs both sporadically and in association with tuberous sclerosis complex (TSC). Sirolimus (rapamycin), an mTORC1 inhibitor, has been shown to stabilize lung function decline and decrease angiomyolipoma tumor size in both TSC and sporadic LAM patients. However, cessation of rapamycin therapy results in recurrent decline in lung function, and regrowth of angiomyolipoma, suggesting that continuous use may be required to maintain its beneficial effects. Recently the investigators have discovered that cyclo-oxygenase (COX) function is altered in cells lacking TSC2, including in a LAM patient-derived angiomyolipoma cell line. COX-2 levels are increased, prostaglandin metabolite levels are increased, and treatment with COX-2 inhibitors are effective in reducing tumor size in two different Tsc mouse models, one a native tumor, and the other a xenograft model. Furthermore, rapamycin does not affect these differences in COX-2 expression or prostaglandin metabolites.

Objectives/Hypothesis: Our preclinical studies indicate that celecoxib (a COX-2 specific inhibitor) decreases the size of TSC2-deficient tumors in Tsc models. Hence the investigators propose this Pilot Clinical Trial to test the safety and tolerability of celecoxib in patients with LAM, with preliminary assessment of potential benefit using multiple approaches.

Specific aims: The primary endpoint of this pilot trial is to test the safety and tolerability of treatment with celecoxib in patients with mild-to-moderate LAM, who are not currently on sirolimus; and to assess the potential benefit of this treatment using the following: 1. Spirometry, 2. MRI measurement of angiomyolipoma size, 3. St. George's Respiratory Questionnaire, 4. VEGF-D serum levels. The investigators will assess Exhaled breath condensate prostaglandin metabolites to confirm effects of celecoxib. The investigators will also develop a novel biomarker of LAM to assess response, quantitative measurement of the number of TSC2 mutant circulating LAM cells, by next generation sequencing.

Study design: The investigators will perform a pilot clinical trial to investigate the safety and tolerability of celecoxib therapy as a single agent for patients with LAM. LAM subjects who are not taking everolimus or rapamycin will be treated with celecoxib at 200mg PO QD for 6 months. They will be monitored for respiratory function and angiomyolipoma size. At the end of the 6 month period, celecoxib will be discontinued, and subjects will be monitored for another 6 months.

Clinical Impact: Sirolimus is the only medical therapy shown to reduce tumor size and stabilize lung function in patients with LAM and TSC-LAM. Although sirolimus has clear benefits, results from the MILES trial suggest that continuous therapy in some form is required, as the rate of decline in lung function resumed when sirolimus was discontinued. The investigators hope that celecoxib will show benefit with minimal toxicity in this trial, and provide an alternative approach for the long term prophylactic/preventive treatment of patients with mild-to-moderate LAM. Our study will include patients with TSC LAM, which often appears to be more slowly progressive than sporadic LAM, and hence long term therapy with celecoxib may have particular benefit in the TSC LAM population. In addition, the investigators will develop a quantitative measure of circulating LAM cell levels as part of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Female of age 18 to 69
* Ability to give informed consent
* Definite diagnosis of LAM Typical cystic change on CT scan of the chest plus one of the following i) biopsy or cytology of any tissue demonstrating LAM, ii) angiomyolipoma, chylothorax, clinical or genetic diagnosis of tuberous sclerosis, iii) serum VEGF-D > 800pg/ml
* post-bronchodilator forced expiratory volume in one second ≥ 70% of predicted and DLCO ≥ 70% predicted during baseline visit.
* Women of childbearing potential must agree to use two forms of barrier contraception after screening visit, for the duration of study participation and for 30 days after last dose.

Exclusion Criteria:

* History of intolerance to non-steroidal anti-inflammatory drugs (NSAIDs)
* History of current regular use (daily most days of the week) of NSAIDs
* History of use of rapamycin or everolimus
* Uncontrolled intercurrent illness
* Pregnant, breast feeding or planning to become pregnant in the next 2 years
* Significant hematological (platelet count <100.000/µl or hepatic abnormalities (Liver function tests >2 times normal).
* Use of an investigational drug within 30 days of study start
* Inability to attend scheduled clinic visits
* Inability to give informed consent
* Inability to perform spirometry
* Creatinine > 1.0 mg/dl or eGFR < 60 ml/min
* Pneumothorax within past 8 weeks
* History of malignancy in the last 2 years other than basal cell skin cancer
* Use of estrogen containing medication within 30 days of enrolment
* Currently taking doxycycline, metformin, lupron or simvastatin
* Unable to undergo MRI
* History of seizure within the last year
* History of hepatitis or known active hepatitis B or C, or HIV positive serology
* Angiomyolipoma of diameter > 4 cm
* History of vascular disease, including myocardial infarction or stroke
* History of ulcers or GI bleeding
* Allergy to sulfonamides, unless subject has previously used Celocoxib without any adverse reactions.
* Age older than 70

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-15; Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Kwiatkowski, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] El-Chemaly S, Taveira-DaSilva A, Bagwe S, Klonowska K, Machado T, Lamattina AM, Goldberg HJ, Jones AM, Julien-Williams P, Maurer R, Rosas IO, Henske EP, Moss J, Kwiatkowski DJ. Celecoxib in lymphangioleiomyomatosis: results of a phase I clinical trial. Eur Respir J. 2020 May 27;55(5):1902370. doi: 10.1183/13993003.02370-2019. Print 2020 May. No abstract available. PMID 32060062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Celecoxib
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Celecoxib
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48 [39 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability in LAM patients
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 12
Participants | 11

2. Secondary Outcome: FEV1
Description: Forced expiratory volume in 1 second
Time Frame: 1 year
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | Celecoxib
Number analyzed (Participants) | 12
ml | 2583 (166)

3. Secondary Outcome: Angiomyolipoma Size Measured Volumetrically on MRI
Description: We are reporting the number of participants in this trial who had angiomyolipoma either at the beginning or end of the study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 12
Participants | 3

4. Secondary Outcome: St. George's Respiratory Questionnaire
Description: St. George's Respiratory Questionnaire is a commonly used questionnaire to assess the respiratory function of an individual.
  The minimum and maximyum socres on this Questionnaire are: 0 and 100. A higher score shows more limitations, so a lower score is better in terms of respiratory function.
  There are no subscales. Below we are providing mean scores for all 9 participants in this trial.
Time Frame: 1 year
Population: Nine of 12 patients who enrolled on the study stayed on study until the end
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib
Number analyzed (Participants) | 9
score on a scale | 20.2 (4.9)

5. Secondary Outcome: VEGF-D Serum Levels
Description: VEGF-D serum levels
Time Frame: 6 months
Population: those who stayed on study until the end
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Celecoxib
Number analyzed (Participants) | 9
pg/mL | 656 [279 to 1865]

6. Secondary Outcome: EBC Prostaglandin Metabolites
Description: We had intended to perform Exhaled breath condensate prostaglandin metabolites. However, this proved to be impossible, and no data was obtained.
Time Frame: 1 year
Arm/Group | Celecoxib
Number analyzed (Participants) | 0

7. Secondary Outcome: Circ LAM Cell Count
Description: We had planned to determine a circulating LAM cell count. However, this proved to be impossible. Therefore, no data was collected.
Time Frame: 1 year
Population: all participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: same as that used by clinicaltrials.gov
Arm/Group | Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=12)
abdominal pain (Gastrointestinal disorders) | 3 (6) — stomach/abdominal pain
headache (Nervous system disorders) | 3 (6)
fatigue (General disorders) | 3 (3) — fatigue
malaise (General disorders) | 2 (2) — malaise

LIMITATIONS AND CAVEATS:
pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT02484664/Prot_SAP_000.pdf